CLINICAL TRIAL: NCT01226472
Title: Open-Label Extension Study of Anti-CCR4 Monoclonal Antibody KW-0761 as Monotherapy in Subjects Who Relapsed After Complete Response on Study KW-0761-001
Brief Title: Extension Study in Subjects Who Relapsed After Complete Response on Study KW-0761-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Collaborators: Kyowa Hakko Kirin Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KW-0761-002
Record Dates: First submitted 2010-10-19; First posted 2010-10-22 (Estimated); Results first posted 2020-12-29 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Peripheral T-cell Lymphoma; Cutaneous T-cell Lymphoma
Keywords: PTCL; CTCL; MF; SS
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous | interventions — mogamulizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- KW-0761 (Experimental)
  Interventions: Biological: KW-0761

INTERVENTIONS:
Biological: KW-0761 — In the first treatment course KW-0761 will be administered i.v. once a week for four weeks, followed by a 2-week observation period. Subsequent treatment courses are permissible for subjects demonstrating a response or maintaining stable disease and will consist of an infusion of KW-0761 every other week.

SUMMARY:
This study will enroll subjects with either Peripheral T-Cell Lymphoma (PTCL) or Cutaneous T-Cell Lymphoma(CTCL),including mycosis fungoides (MF) and Sezary Syndrome (SS), who have relapsed after achieving a complete response in study, KW-0761-001.

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject has relapsed after achieving a complete response to treatment with KW 0761 for PTCL or CTCL on study, KW-0761-001.

  2. The subject has an Eastern Cooperative Oncology Group (ECOG) performance status score of < 2 at study entry.

  3. The subject is >18 years of age. 4. The subject has adequate hematological function: absolute neutrophil count [ANC] >1,500 cells/uL and platelets >100,000 cells/uL,except in patients with known bone marrow involvement where absolute neutrophil count [ANC] must be > 1,000 cells/uL and platelets >75,000 cells/uL.

  5. The subject has adequate hepatic function: bilirubin ≤ 1.5 times the specific institutional upper limit of normal [ULN]; aspartate transaminase [AST] and alanine transaminase [ALT] each ≤ 2.5 x ULN or ≤ 5.0 x ULN in the presence of known hepatic malignancy.

  6. The subject has serum creatinine ≤1.5 x ULN or a calculated creatinine clearance >60 mL/min.

  7. Subjects with MF and a history of staphylococcus colonization are eligible provided they continue to receive stable doses of prophylactic antibiotics.

Exclusion Criteria:

1. The subject has received any type of treatment for their disease since completing study, KW-0761-001.
2. The subject has a significant uncontrolled intercurrent illness including, but not limited to: uncontrolled infection requiring antibiotics; clinically significant cardiac disease (class III or IV of the New York Heart Association [NYHA] classification); unstable angina pectoris; angioplasty, stenting, or myocardial infarction within 6 months; uncontrolled hypertension (systolic blood pressure >160 mmHg, diastolic BP >100 mmHg, found on two consecutive measurements separated by a 1 week period) despite two anti-hypertensive medications; clinically significant cardiac arrhythmia; or uncontrolled diabetes.
3. Subjects on any immunomodulatory drug, (other than low dose corticosteroids equivalent to a daily dose of 10 mg of prednisone
4. The subject has a psychiatric illness, disability or social situation that would compromise the subject's safety or ability to provide consent, or limit his or her compliance with study requirements.
5. The subject has experienced allergic reactions to monoclonal antibodies or other therapeutic proteins.
6. Subjects with active herpes simplex or herpes zoster.
7. Subjects with known autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-08; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Kurman, M.D., Study Director — Kyowa Hakko Kirin Pharma, Inc.
Locations (1):
- Stanford University, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | KW-0761
Started | 1
Completed | 0
Not Completed | 1
Not completed — Progressive Disease | 1

BASELINE CHARACTERISTICS:
Population: Only subjects with PTCL or CTCL who subsequently relapsed after achieving a CR in Study KW 0761-001 and who provided signed informed consent were eligible to enroll in the study.
Arm/Group | KW-0761
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Hispanic or Latino | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Global Composite Response (Skin, Blood, Lymph Nodes)as Determined by Skin Evaluations, Blood Counts and PET/CT Imaging
Time Frame: one year
Population: Safety Analysis Set: All subjects who received at least one dose of KW-0761 (even a partial dose).
Measure: Number; unit: days
Arm/Group | KW-0761
Number analyzed (Participants) | 1
days
  Progression-Free Survival (PFS) | 260
  Time to Progression (TTP) | 260
  Duration of Overall Response (DR) | 232

2. Secondary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability.
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | KW-0761
Number analyzed (Participants) | 1
Participants
  With Any TEAE | 1
  With Any Drug-related TEAE | 0
  With Any TEAE with an Outcome of Death | 0
  With Any Serious TEAE | 0
  With Any Drug-related Serious TEAE | 0
  With Any Serious TEAE with an Outcome of Death | 0

ADVERSE EVENTS:
Arm/Group | KW-0761
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KW-0761 (N=1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days